CLINICAL TRIAL: NCT05401669
Title: Transradial Versus Transfemoral Access for Cerebral Angiography
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Yuxiang Gu, Vice-president of Huashan Hospital west campus, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021Y9308
Record Dates: First submitted 2022-05-23; First posted 2022-06-02 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Angiography
Keywords: Cerebral Angiography; Transfemoral Arterial access; Transradial Arterial access

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trans-radial artery access (Experimental)
  Interventions: Procedure: Trans-radial access
- Trans-femoral Artery access (Active Comparator)
  Interventions: Procedure: Trans-femoral access

INTERVENTIONS:
Procedure: Trans-radial access — Cerebral angiography performed by trans-radial access
  Arms: Trans-radial artery access
Procedure: Trans-femoral access — Cerebral angiography performed by trans-femoral access
  Arms: Trans-femoral Artery access

SUMMARY:
This study is multi-center, prospective, randomized (1:1) controlled trial designed to assess and compare the feasibility, safety and success of Transradial access (TRA) versus Transfemoral access (TFA) for diagnostic cerebral angiography.

DETAILED DESCRIPTION:
TFA is traditional approach for diagnostic cerebral angiography, which has several limitations and complications including pain and discomfort, retroperitoneal hemorrhage, pulmonary embolism and increased admissions. Transradial coronary angiography has demonstrated preponderance to circumvent this limitations and complications. However, this has not been studied in cerebral angiography. So, the purpose of this study is to assess and compare the feasibility, safety and success of TRA versus TFA for diagnostic cerebral angiography.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years old;
2. Scheduled to undergo diagnostic cerebral angiography;
3. Suitable for cerebral angiography via TRA and TFA access, with a radial artery diameter ≥2mm confirmed by ultrasonography;
4. Modified Rankin Scale (mRS) score ≤2;
5. Provided written informed consent.

Exclusion Criteria:

1. Severe stenosis of the radial, brachial, subclavian, brachiocephalic, iliac or common femoral arteries, or any significant vascular disease (such as aortic aneurysm, etc.) that may obstruct guidewire passage;
2. Arteriovenous fistula for hemodialysis present in the right upper limb;
3. Planned interventional surgery within 24 hours of the initial study angiography;
4. Requirement for cerebral angiography in an emergency department;
5. Use of general anesthesia;
6. Any contraindication to cerebral angiography, such as allergy or intolerance to the contrast media, uncorrected severe coagulation disorders, arterial dissection in the target vessel, puncture site infection, or renal insufficiency (Creatinine [Gr] > 3 times of the upper limit of normal [ULN]), etc.;
7. Women who are pregnant or planning to become pregnant within 1 year;
8. Participation in another clinical trial;
9. Any other condition deemed unsuitable for participation by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 748 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
the rate of successful diagnostic cerebral angiography | 24 hours
  the successful superselection of the aortic arch vessel without changing the arterial approach, with angiography results meeting diagnostic requirements

SECONDARY OUTCOMES:
the rate of successful accurate diagnosis | 24 hours
the duration of angiography | During procedure
  time taken to do the full procedure
the duration of fluoroscopy | During procedure
  Radiation time (min) after placing the sheath at the initial puncture site until the completion of the diagnostic cerebral angiography
the bedridden time | 24 hours
the Visual Analogue Scale (VAS) score | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yuxiang Gu, PhD,MD, Study Chair — department of Neurosurgery, Huashan Hospital,Fudan University; Wei Ni, PhD,MD, Study Director — department of Neurosurgery, Huashan Hospital,Fudan University
Locations (1):
- Huashan Hospital, Shanghai, Shangai, China

IPD SHARING:
Plan to Share IPD: No